CLINICAL TRIAL: NCT05202561
Title: A Single-Arm, Open-Label, Exploratory Study to Evaluate the Safety of RNA Tumor Vaccine Injection Alone/in Combination With PD-1 Inhibitor in the Treatment of Advanced Solid Tumors With KRAS Mutation
Brief Title: A Study of RNA Tumor Vaccine in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Principal Investigator, Wang Zishu, MD, The First Affiliated Hospital of Bengbu Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LWY21084CBY
Record Dates: First submitted 2022-01-19; First posted 2022-01-21 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Advanced Solid Tumor
Keywords: KRAS mutation; RNA tumor vaccine; injection; PD-1; immunotherapy; Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Drug: RNA tumor vaccine Administration: intramuscular injection Dose: 600 ng/ time Dosing cycle: Day 1, day 4, day 7, and day 14.
  Interventions: Biological: RNA tumor vaccine
- Arm B (Experimental): Drug: RNA tumor vaccine+Navuliumab Administration: intravenous injection Dose: 3 mg/kg Timing of administration: Administration was initiated 14 days after the first intramuscular injection of the RNA tumor vaccine.
  Duration of administration: once every 2 weeks.
  Interventions: Biological: RNA tumor vaccine+Navuliumab

INTERVENTIONS:
Biological: RNA tumor vaccine — Subjects will receive single dose of RNA tumor vaccine injection on day 1, day 4, day 7, and day 14, each dose of 600 ng.
  Arms: Arm A
Biological: RNA tumor vaccine+Navuliumab — RNA tumor vaccine+Navuliumab Subjects will receive maintenance therapy with a PD-1 inhibitor in addition to monotherapy with the RNA tumor vaccine injection. Subjects received a single dose of RNA vaccine injection on day 1, day 4, day 7, and day 14, with each dose of 600 ng. Inhibitors, accept the Navuliumab on day 14, the recommended dose is 3 mg/kg, intravenous injection every 2 weeks.
  Arms: Arm B

SUMMARY:
This is a single-arm, open-label, clinical pharmacology study to evaluate the safety of RNA tumor vaccine injection alone/in combination with PD-1 inhibitor in the treatment of advanced solid tumors with KRAS mutation.

The purpose of this study is to evaluate the safety and tolerability, antitumor activity, The immunoreactivity, pharmacokinetics and of RNA tumor vaccine.

DETAILED DESCRIPTION:
This is an investigator initiated , sinle-arm, open-label clinical pharmacology to evaluate the safety and efficacy of RNA vaccine injection alone/in combination with PD-1 inhibitor in patients with advanced solid tumors with KRAS mutation (G12C, G12D, or G12V) and HLA type HLA-A11:01 or HLA C08:02. 10 subjects were enrolled. Monotherapy and combination therapy are included. Some eligible subjects will receive single drug therapy with RNA tumor vaccine injection, and some will receive combined treatment with PD-1. Among them:

Arm A:RNA tumor vaccine The single-agent study evaluated the safety, efficacy and pharmacokinetic characteristics of a fixed-dose (600ng) KRAS-targeted RNA vaccine injection as a single agent in humans. Eligible subjects will receive a single dose of RNA vaccine injection on day 1, day 4, day 7, and day 14, each dose of 600ng.

Arm B: RNA tumor vaccine+Navuliumab Subjects will receive maintenance therapy with a PD-1 inhibitor in addition to monotherapy with the RNA tumor vaccine injection. Subjects received a single dose of RNA vaccine injection on day 1, day 4, day 7, and day 14, with each dose of 600 ng. Inhibitors, accept the Navuliumab on day 14, the recommended dose is 3 mg/kg, intravenous injection every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is at least 18 years old with no gender limitation;
2. Patients with advanced malignant solid tumors confirmed by histopathology or cytology and failed to receive standard treatment or without standard treatment;
3. Identification of at least one KRAS mutation: G12C, G12D or G12V;
4. The subtype was identified as HLA-A11:01 or C08:02;
5. Have at least one measurable lesion according to RECIST V1.1;
6. ECOG PS score was 0-2 in the Eastern Oncology Group;
7. Full organ and bone marrow function, as defined below:
8. Sign written informed consent and be able to comply with the visits and related procedures specified in the program;
9. Eligible fertile patients (male and female) must agree to use a reliable contraceptive method (hormonal or barrier methods or abstinence) during the study period;

Exclusion Criteria:

1. A history of severe allergy to biological products;
2. Those in pregnancy or lactation;
3. The expected survival time is less than 3 months;
4. Those who have undergone major surgery within 4 weeks prior to signing the informed consent, or who plan to undergo major surgery during the study period;
5. Received chemotherapy, biotherapy, endocrine therapy, immunotherapy and other anti-tumor drugs within 2 weeks before the first administration;
6. Participating in other clinical studies;
7. Patients with central nervous system metastasis or a history of central nervous system metastasis;
8. Adverse effects of previous antitumor therapy have not recovered to NCI CTCAE V5.0 rating ≤1 (except hair loss);
9. Serious cardiovascular and cerebrovascular diseases, hypertension that is still poorly controlled after standard treatment (systolic blood pressure > 150mmHg, diastolic blood pressure > 90mmHg);
10. Patients with active ulcers and gastrointestinal bleeding;
11. Patients with uncontrollable pleural effusion, abdominal effusion and pericardial effusion;
12. Active infection requiring treatment;
13. HIV, HCV, syphilis, CMV, EBV infected patients; Patients with active HBV replication;
14. A history of interstitial lung disease;
15. The patient has an autoimmune disease or is in an immunosuppressed state; Current systemic steroid use (except recent or current inhaled steroid use);
16. Other conditions that the investigator assessed as ineligible for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-01-19 (Estimated); Study Completion 2024-01-19 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 months
  Graded according to the NCI CTCAE version 5.0.

SECONDARY OUTCOMES:
To evaluate the antitumor activity | Up to 2 years
  To assess per RECIST and iRECIST
The changes of the immunoreactivity during treatment. | Up to 28 Days
  Peripheral blood T lymphocyte subtype

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital Bengbu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No